CLINICAL TRIAL: NCT04118556
Title: A Multicenter, Open-label, Randomized, Phase I/II Clinical Trial Comparing Safety and Durable Overall Response Day 56 in Patients With Steroid Resistent Acute GvHD After Allogeneic Hematopoietic Stem Cell Transplant Treated With DSC or BAT
Brief Title: Decidua Stroma Cells for Steroid Resistent Acute Graft-versus-host Disease After Allo-HSCT
Acronym: 2017-00355
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mats Remberger (Other)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Sponsor-Investigator, Mats Remberger, Professor, Uppsala University Hospital
Organization: Uppsala University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSC-BROMS-1; 2019-002186-36 (EudraCT Number)
Record Dates: First submitted 2019-09-27; First posted 2019-10-08 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: GVHD, Acute
Keywords: DSC; BAT; GVHD; HSCT
MeSH Terms: conditions — Graft vs Host Disease | interventions — Eosinophil Cationic Protein; Everolimus; Sirolimus; Etanercept; vedolizumab; ruxolitinib; Infliximab

STUDY DESIGN:
Intervention Model Description: A randomized (1:1) phase II open label study of DSC compared to Investigator choice Best Available Therapy (BAT) in allogeneic hematopoietic stem cell transplant recipients with Grades II-IV steroid refractory acute graft vs. host disease. Patients will receive 2 doses of DSC. Additional doses (up to 4 doses) may be given depending on response.
  No cross-over are planned in the second stage of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decidua Stroma Cells (DSC) (Experimental): Placenta derived decidua stroma cells (DSC). In the first phase I part, two different dose levels will be used, 1x10^6/kg and 3x10^6/kg. Two doses, one week apart, will be given. The decision to proceed to the next dose level will depend on results observed at the previous dose level.
  The dose in the randomized part will be based on the findings in the phase I part. In the Phase II study all patients will receive 2 doses, one week apart. Depending on response, up to 6 doses in total may be given. Additional doses (beyond the first 2 doses) may be given one week apart until response.
  Interventions: Biological: Decidua Stroma Cells (DSC)
- Best Available Treatment (BAT) (Active Comparator): The BAT in this study will freely be identified by the Investigator prior to patient randomization and may include treatments such as: anti-thymocyte globulin (ATG), extracorporeal photopheresis (ECP), low-dose methotrexate (MTX), mycophenolate mofetil (MMF), mTOR inhibitors (everolimus or sirolimus), etanercept, vedolizumab, ruxolitinib or infliximab. Dose and frequency will depend on label (where approved) and institutional guidelines for various BAT.
  Interventions: Drug: Best available Treatment (BAT)

INTERVENTIONS:
Biological: Decidua Stroma Cells (DSC) — Placenta-derived Decidua Stroma Cells. The product consists of a viable allogeneic DSCs frozen in 5% of human serum albumin (HSA) in sodium chloride (NaCl) 0.9% and 10% dimethylsulfoxide (DMSO), that is thawed and immediately diluted in 40 mL sodium chloride (NaCl) 0.9% prior to infusion. That will give a final concentration of 2.2% HSA and 2% DMSO.
  DSC will be infused when steroid-refractory acute GVHD after allogenic stem-cell transplantation has been diagnosed. Two doses, one week apart, will be given to all patients. Additional doses will be used depending on response.
  Arms: Decidua Stroma Cells (DSC)
Drug: Best available Treatment (BAT) — The BAT in this study will freely be identified by the Investigator prior to patient randomization and may include treatments such as: extracorporeal photopheresis (ECP), low-dose methotrexate (MTX), mycophenolate mofetil (MMF), mTOR inhibitors (everolimus or sirolimus), etanercept, vedolizumab, ruxolitinib or infliximab. Dose and frequency will depend on label (where approved) and institutional guidelines for various BAT.
  Other Names: ECP, Everolimus, Sirolimus, Etanercept, Vedolizumab, Ruxolitinib, Infliximab.
  Arms: Best Available Treatment (BAT)

SUMMARY:
A randomized (1:1) phase II open label study of DSC compared to Investigator choice Best Available Therapy (BAT) in allogeneic hematopoietic stem cell transplant recipients with Grades II-IV steroid refractory acute graft vs. host disease in the second part of the study. Patients will receive 2 doses of DSC. Additional doses (up to 4 doses) may be given depending on response.

No cross-over are planned in the second stage of the study.

DETAILED DESCRIPTION:
Main inclusion criteria:

Adult patients (age ≥ 18 years) with steroid refractory (SR) acute GvHD (aGVHD) grades II-IV after allo-HSCT.

Signed written study informed consent once SR-aGvHD is confirmed.

Main exclusion criteria:

Presence of an active uncontrolled infection requiring treatment. Has received systemic treatment for aGvHD apart from steroids. Clinical presentation resembling de novo chronic GvHD or GvHD overlap syndrome. Known human immunodeficiency virus infection (HIV). Patients suffering on active tuberculosis or viral hepatitis. Significant respiratory disease Presence of severely impaired renal function Patients with coagulopathy Pregnant or nursing (lactating) women Malignancy that has required treatment in the previous two years Any condition that would, in the Investigator's judgment, interfere with full participation in the study.

Design:

The trial is a Phase II, randomized (1:1), open label study investigating the efficacy and safety of DSC vs. BAT added to the patient's immunosuppressive regimen in adults with SR-aGvHD.

The primary objectives will be safety and to compare durable overall response (DOR) at 56 days after randomization between patients receiving DSC with patients receiving BAT as treatment for SR acute GvHD grades II-IV. Target enrollment is 50 patients, 25 in the DSC treatment-arm and 25 in the BAT arm. Patients will be given the optimal dose of DSC from the Phase I, dose escalating part of the study, as mentioned above. At least 2 doses of DSC will be given one week apart. Additional doses of DSC (maximum 4 doses) may be given depending on response. Additional doses (beyond the first 2 doses) may be given one week apart until response, or whenever needed if aGVHD flare occur within 6 months after randomization (EOT).

BAT: Investigator's choice Best Available Therapy (BAT) will vary depending upon Investigator's choice identified prior to randomization. Dose and frequency will depend on label (where approved) and institutional guidelines for various BAT.

Primary objective

* Assess the Safety of DSC.
* Durable Overall Response (DOR) at Day 56.

Secondary objectives

* To assess Overall Response Rate (ORR) at day 28
* To assess 1-year Overall Survival (OS)
* To assess 1-year Non-Relapse Mortality (NRM)
* To assess incidence of infections

Exploratory objectives

* To assess the cumulative steroid dose until Day 56 and Day 90
* To assess Event-Free Survival (EFS)
* To assess incidence of Malignancy Relapse/Progression
* To measure the incidence of chronic GvHD
* To measure immune reconstitution
* To evaluate changes in Patient Reported Outcomes

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (age ≥ 18 years) with steroid refractory acute GvHD grades II-IV after allo-HSCT.
2. Signed written study informed consent once SR-aGvHD is confirmed.

Exclusion Criteria:

1. Presence of an active uncontrolled infection including significant bacterial, fungal, viral or parasitic infection requiring treatment.
2. Has received systemic treatment for aGvHD apart from steroids.
3. Clinical presentation resembling de novo chronic GvHD or GvHD overlap syndrome.
4. Pregnant or lactating women.
5. Significant respiratory disease.
6. Presence of severely impaired renal function
7. Any corticosteroid therapy for indications other than aGvHD
8. Previous participation in a study of any investigational treatment agent within 30 days
9. Known human immunodeficiency virus infection (HIV).
10. Patients suffering on active tuberculosis or viral hepatitis
11. Significant respiratory disease
12. Presence of severely impaired renal or liver function
13. History of progressive multifocal leuko-encephalopathy
14. Patients with coagulopathy
15. History of severe chronic history of heart disease
16. Any condition that would, in the Investigator's judgment, interfere with full participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability evaluation including Severe Adverse Events (SAE). | 5 years
  Adverse events will be assessed and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Durable Response to treatment | 56 days
  Durable Overall Response (DOR) day 56.

SECONDARY OUTCOMES:
Number of patients with overall response (CR+PR) at day 28 | 28 days
  Overall Response Rate (ORR) at day 28.
Rate of Survival | 1 year
  Death within 1 year after inclusion in study.
Incidence of Non-Relapse Mortality (NRM) | 1 year
  Death of any cause with enduring complete remission.
Incidence of infections | 1 year
  Serious infections occurring after inclusion in study.
Change of Quality of Life | 1 year
  Change of self-experienced well-being (Quality of Life)(FACT-BMT version 4) at four time-points after inclusion. Scoring procedures consist of summing the items with reversed scoring (0-4p where 0=best and 4=worst) for several items which produces individual subscale scores (0-24/28p) and an overall score (0-200p).
  The FACT-BMT (Functional Assessment of Cancer Therapy-Bone Marrow Transplant) has a total of 50 questions. This is a questionnaire of general questions divided into four primary quality of life domains: physical well-being (PWB; 7-items), social/family well-being (SWB; 7-items), emotional well-being (EWB; 6-items); and functional well-being (FWB; 7-items), 18 items address the BMT related side effects, specifically designed to assess the BMT patients' quality of life. Five other questions from different QoL questionnaire were added as they were considered relevant to FACT-BMT.
Incidence of Relapse | 5 year
  Recurrence of the disease the patient were transplanted for.
Incidence of secondary malignancies | 5 year
  Occurrence of other malignancies than the patient were transplanted for.
Incidence of chronic GVHD | 5 year
  Occurrence of chronic GVHD.

CONTACTS AND LOCATIONS:
Overall Officials: Mats Remberger, Professor, Study Director — KFUE, Uppsala University Hospital, Uppsala, Sweden; Ulla Olsson-Strömberg, AssProfessor, Principal Investigator — Dep of Hematology, Uppsala University Hospital, Uppsala, Sweden
Locations (6):
- Copenhagen Univerity Hospital, Copenhagen, Denmark
- Oslo University Hospital, Oslo, Norway
- Sweden (4):
  - Gothenburg University Hospital, Gothenburg
  - Lund University Hospital, Lund
  - Karolinska University Hospital, Stockholm
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ringden O, Baygan A, Remberger M, Gustafsson B, Winiarski J, Khoein B, Moll G, Klingspor L, Westgren M, Sadeghi B. Placenta-Derived Decidua Stromal Cells for Treatment of Severe Acute Graft-Versus-Host Disease. Stem Cells Transl Med. 2018 Apr;7(4):325-331. doi: 10.1002/sctm.17-0167. Epub 2018 Mar 13. PMID 29533533
- [Result] Sadeghi B, Remberger M, Gustafsson B, Winiarski J, Moretti G, Khoein B, Klingspor L, Westgren M, Mattsson J, Ringden O. Long-Term Follow-Up of a Pilot Study Using Placenta-Derived Decidua Stromal Cells for Severe Acute Graft-versus-Host Disease. Biol Blood Marrow Transplant. 2019 Oct;25(10):1965-1969. doi: 10.1016/j.bbmt.2019.05.034. Epub 2019 Jun 4. PMID 31173898